CLINICAL TRIAL: NCT00204776
Title: A Phase II Trial of Capecitabine and Oxaliplatin in Metastatic Breast Cancer
Brief Title: XELOX for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CO04104; 2004-0340
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine and Oxaliplatin

SUMMARY:
Both capecitabine and oxaliplatin have single agent activity in breast cancer. The combination has improved activity in other solid tumors. This study seeks to assess the activity of the combination in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* preserved organ function
* good performance status
* no more than one prior therapy
* no active brain metastasis

Exclusion Criteria:

* No prior capecitabine or oxaliplatin
* no con-current therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2005-03; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Toxicity
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Morgan-Meadows, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States